CLINICAL TRIAL: NCT06264284
Title: Emergency (Red Code) Cesarean Section : Maternal and Fetal Prognosis Depending on Anesthetic Modalities in a Level 3 Maternity Ward
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, STANOWSKI Mattieu, MD, Central Hospital, Nancy, France
Other Study IDs: 2023PI163
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia Complication
Keywords: c-section, cesarean section, epidural anesthesia, anesthesia complication
MeSH Terms: interventions — Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epidural anesthesia
  Interventions: Procedure: epidural anesthesia
- general anesthesia
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: epidural anesthesia — Emergency cesarean section (red code) with epidural anesthesia
  Groups: epidural anesthesia
Procedure: general anesthesia — Emergency cesarean section (red code) with general anesthesia
  Groups: general anesthesia

SUMMARY:
We try to evaluate whether the type of anesthesia used influences the occurrence of perioperative maternal complications as well as neonatal outcome on emergency (Red Code) Cesarean Section.

This study occurred in a Level 3 Maternity Ward.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* emergency "code red" cesarean section

Exclusion Criteria:

* Any other intervention
* Planned cesarean section

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who have undergone an emergency "code red" cesarean from July 19, 2018 to July 19, 2023, at the Nancy CHRU maternity ward
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
To evaluate whether the type of anesthesia used influences the occurrence of perioperative maternal complications as well as neonatal outcome | From July 19, 2018 to July 19, 2023.
  Identify all pregnant women who received an emergency "code red" cesarean section
  Confront epidural anesthesia and general anesthesia on maternal complications (low blood pressure, anesthetic failure) and neonatal outcomes (Apgar scores, arterial pH at the umbilical cord, arterial lactate, need for tracheal intubation at birth, admission of the newborn to intensive care/intensive care, death)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanowski, Nancy, France